CLINICAL TRIAL: NCT04282941
Title: Phase III Clinical Trial, Randomized, Multicentre, Double Blind to Evaluate Two Guidelines for the Administration of Ibuprofen in the Treatment of Persistent Ductus Arteriosus Eco-guided: Impact in the Intestinal Prognosis
Brief Title: Clinical Trial to Evaluate Two Guidelines for the Administration of Ibuprofen in the Treatment of Persistent Ductus Arteriosus Eco-guided: Impact in the Intestinal Prognosis
Acronym: IBU24h-EchoG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-002974-11
Record Dates: First submitted 2020-02-05; First posted 2020-02-25 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-07

CONDITIONS: Persistent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Ibuprofen; Infusions, Intravenous

STUDY DESIGN:
Intervention Model Description: Administration schedule A: Ibuprofen in continuous iv infusion and EchoG. Each cycle will be 3 doses.
  Administration schedule B: slow iv bolus Ibuprofen and EchoG. Each cycle will be 3 doses.
Who Masked: Participant, Investigator
Masking Description: A randomized system with closed envelopes will be designed in which patients will be assigned to one of the 2 treatment groups, stratified by gestational age (<28 weeks and ≥28 weeks) and by hospital center. In each center and each stratum, they will be randomly assigned in a 1: 1 ratio to each group of study. The assignment will be sequential.
  The doctors responsible for the patient will be blind to the intervention but will be responsible for the sealed envelopes, and at the time of patient randomization, will deliver the sealed envelope corresponding to the nurses responsible for the preparation of the medication.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen in continuous (24 hours) iv infusion and EchoG (Experimental): The first dose of ibuprofen will be 10 mg / kg to be administered as a continuous infusion for 24 hours. An echocardiogram will be performed before each of the following 2 doses of 5 mg / Kg and will only be administered if it meets echocardiographic criteria that indicate open DA (observation of ductus permeability with color Doppler regardless of its size). Each dose will be administered as a 24-hour continuous infusion.
  Interventions: Drug: Ibuprofen in continuous (24 hours) iv infusion and EchoG
- IV bolus Ibuprofen slow (15 minutes) and EchoG (Experimental): The first dose of ibuprofen of 10 mg / Kg to be administered in slow iv bolus (15 minutes). Before each of the following 2 doses of 5 mg / Kg, echocardiography will be performed and will only be administered if it meets the echocardiographic criteria indicated by open DA (observation of ductus permeability in color Doppler regardless of its size). Each dose will be administered in iv boluses in 15 minutes
  Interventions: Drug: IV bolus Ibuprofen slow (15 minutes) and EchoG

INTERVENTIONS:
Drug: Ibuprofen in continuous (24 hours) iv infusion and EchoG — The first dose of ibuprofen will be 10 mg / kg to be administered as a continuous infusion for 24 hours. An echocardiogram will be performed before each of the following 2 doses of 5 mg / Kg and will only be administered if it meets echocardiographic criteria that indicate open DA (observation of ductus permeability with color Doppler regardless of its size). Each dose will be administered as a 24-hour continuous infusion.
  Arms: Ibuprofen in continuous (24 hours) iv infusion and EchoG
Drug: IV bolus Ibuprofen slow (15 minutes) and EchoG — The first dose of ibuprofen of 10 mg / Kg to be administered in slow iv bolus (15 minutes). Before each of the following 2 doses of 5 mg / Kg, echocardiography will be performed and will only be administered if it meets the echocardiographic criteria indicated by open DA (observation of ductus permeability in color Doppler regardless of its size). Each dose will be administered in iv boluses in 15 minutes
  Arms: IV bolus Ibuprofen slow (15 minutes) and EchoG

SUMMARY:
Persistent ductus arteriosus (DA) is a common entity in the premature newborn and is associated with high morbidity and mortality. There is still controversy about which is the best treatment for its closure. Children with AD who receive pharmacological treatment present more frequently than other premature children, necrotizing enterocolitis or isolated intestinal perforation.

At the present time, the conventional treatment of DA consists in the administration of intravenous ibuprofen, slow bolus in 3 daily doses 10-5-5 mg / kg / day. Recently, it has been observed that treatment with ibuprofen in continuous iv infusion for 3 days seems to be more effective in closing DA than conventional treatment for 3 days with the same dose but in slow iv bolus. This experimental treatment reduced the incidence of associated necrotizing enterocolitis. Our group demonstrated in a previous pilot trial that the guided treatment with echocardiography (EchoG) of DA with ibuprofen compared with conventional treatment, allows to reduce the number of doses to the patient. The EchoG treatment thus presents a potential reduction of side effects associated with medication, this resulted in a tendency to have a lower incidence of necrotising enterocolitis in the experimental group. This multicenter clinical trial aims to test the hypothesis that the combination of 2 experimental treatments, the use of ibuprofen in continuous perfusion and EchoG, reduces the incidence of digestive side effects (necrotising enterocolitis or isolated intestinal perforation) compared to the treatment also guided by echocardiography but slow bolus iv.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with less 33 weeks of gestational age
* DA ≥ 1.5 mm with decision to start pharmacological treatment
* Informed consent signed by the legal representative

Exclusion Criteria:

* Consent denied
* Presence of serious congenital alterations
* Congenital heart disease
* Contraindication for the administration of IB: oligoanuria (diuresis <1cc / kg / h), bleeding severe recent intraventricular (HIV grade III or extensive periventricular hemorrhagic infarction), serum creatinine> 1.5 mg / dl or clinical suspicion of intestinal ischemia.

Ages: 0 Minutes to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Change the incidence of necrotizing enterocolitis or isolated intestinal perforation in preterm infants receiving treatment for closure of AD with ibuprofen in continuous IV perfusion and EchoG vs iv and EchoG boluses | 40 weeks
  Change the incidence of necrotizing enterocolitis or isolated intestinal perforation in preterm infants receiving treatment for closure of AD with ibuprofen in continuous IV perfusion and EchoG vs iv and EchoG boluses

SECONDARY OUTCOMES:
To Identify genetic polymorphisms asociated to refractory medical treatment of AD and in those most vulnerable to presenting necrotizing enterocolitis or isolated intestinal perforation. | Day 0(Visit 1)
  Identify genetic polymorphisms in patients refractory to medical treatment of AD and in those most vulnerable to presenting necrotizing enterocolitis or isolated intestinal perforation.

OTHER OUTCOMES:
To Assess the incidence of neonatal morbidity associated with each of the forms of treatment | up to 40 Weeks Postmenstrual age
  Assess the incidence of neonatal morbidity associated with each of the forms of treatment
To Assess the neonatal mortality associated with each of the forms of treatment | up to 40 Weeks Postmenstrual age
  Assess the neonatal mortality associated with each of the forms of treatment

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitario La Paz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Quirón Salud Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Undecided